CLINICAL TRIAL: NCT07092657
Title: Effectiveness of an Educational Intervention of Spirituality in Nursing Professionals Working in Critical Health Care Settings to Promote Spiritual Self-care.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ECA01122024
Record Dates: First submitted 2025-06-19; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Spirituality; Nursing; Intensive Care (ICU)
Keywords: Spirituality; Critical care nursing; Nursing care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention under study, neither the participants nor the professional who will carry out the intervention can be masked. Therefore, masking will be done in the following way: a) the intervention provider will not know the outcome indicators of the study, b) the outcome evaluator will not know to which group (intervention or control) the participants will belong.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participant group/arm (Experimental): Educational and behavioral nursing intervention, created to strengthen the spiritual perspective of nursing professionals acting in critical care settings and improve their professional practice by favoring their spiritual self-care.
  Interventions: Other: Nursing Education Intervention
- Control: conventional attention (No Intervention): The control group will receive a single educational session on spiritual management guidelines.

INTERVENTIONS:
Other: Nursing Education Intervention — Four standardized sessions. With a duration of 40 to 60 minutes each session, once a week for a period of one month and a follow-up one month after the end of the intervention. Interventions are carried out at different times depending on the availability of the nursing professionals.
  Arms: Participant group/arm

SUMMARY:
This study will evaluate the effect of an educational intervention of spirituality in nursing professionals acting in critical care contexts to favor spiritual self-care, compared with the conventional care group. The educational intervention adopts Pamela Reed's theory of the transcendence of the self as a theoretical reference, which facilitates the understanding of the phenomenon of spirituality by adopting an integral approach focused on personal growth. To determine the effect of the intervention, the Spiritual Perspective Scale (SPS) developed by Reed will be applied.

DETAILED DESCRIPTION:
Since its historical origins, nursing has been deeply linked to values and principles that give it a solid spiritual heritage. This spiritual connection has been the basis on which the profession has developed, allowing it to evolve without losing its fundamental essence.

In contexts of high emotional demand, such as critical care environments, professionals are faced with multiple spiritual needs that produce existential crises in the search for meaning and purpose, then spirituality acts as a source of strength that not only helps to face challenges, but also promotes greater satisfaction in their daily work.

Thus, the integration of spirituality in the workplace has demonstrated multiple benefits such as increased motivation and commitment, greater job satisfaction and significant improvements in mental and emotional health.

ELIGIBILITY:
Inclusion Criteria:

* Work in a critical unit of the institutions where the study will be carried out.
* Have a minimum experience of 6 continuous months in critical care contexts.
* Have a score of 35-45 points (moderate) and 10-30 points (low).

Exclusion Criteria:

* Nursing professional who fails to complete full participation in the study (pre- test, nursing intervention and post-test).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Spiritual perspective | 2 mounths
  The final average score of each participant on the Spiritual Perspective Scale at the end of the intervention and one month after its completion. The scale consists of 10 items that measure spiritual beliefs and behaviors using a 6-point Likert scale for a score ranging from 10 to 60, classifying values as low spirituality from 10 to 30 points, moderate spirituality from 31 to 45 points, and high spirituality from 46 to 60 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Antioquia, Facultad de Enfermería, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtgoz A, Keten Edis E, Erarslan R. Spiritual Care Competencies and the Frequency of Spiritual Care Practices of Nurses in Turkey. J Relig Health. 2024 Jun;63(3):1747-1760. doi: 10.1007/s10943-023-01884-7. Epub 2023 Aug 4. PMID 37540306
- [Background] Torres-Contreras CC, Vargas-Escobar LM, Triana-Rodriguez JY, Canon-Montanez W. [Spiritual Care Competence in Nursing: Integrative Literature ReviewCompetencia no cuidado espiritual em enfermagem: revisao integrativa da literatura]. Rev Cuid. 2023 Sep 3;14(2):e06. doi: 10.15649/cuidarte.2635. eCollection 2023 May-Aug. Spanish. PMID 40115201
- [Background] Wu X, Hayter M, Lee AJ, Yuan Y, Li S, Bi Y, Zhang L, Cao C, Gong W, Zhang Y. Positive spiritual climate supports transformational leadership as means to reduce nursing burnout and intent to leave. J Nurs Manag. 2020 May;28(4):804-813. doi: 10.1111/jonm.12994. Epub 2020 Mar 25. PMID 32145113
- [Background] Atarhim MA, Lee S, Copnell B. An Exploratory Study of Spirituality and Spiritual Care Among Malaysian Nurses. J Relig Health. 2019 Feb;58(1):180-194. doi: 10.1007/s10943-018-0624-0. PMID 29679189
- [Background] Abdollahyar A, Baniasadi H, Doustmohammadi MM, Sheikhbardesiri H, Yarmohammadian MH. Attitudes of Iranian Nurses Toward Spirituality and Spiritual Care. J Christ Nurs. 2019 Jan/Mar;36(1):E11-E16. doi: 10.1097/CNJ.0000000000000581. PMID 30531521